CLINICAL TRIAL: NCT03662646
Title: Clock Gene Disruption May be an Initial Manifestation of IBD and Celiac .
Brief Title: Circadian Rhythms in Patients With IBD or Celiac Disease Upon Diagnosis and Medical Follow-up
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Dr. Yael Weintraub, Prof. Shlomi Cohen, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMAC-16-YW-0200-CTIL
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Bowel Diseases; Circadian Dysregulation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood, stool and intestinal mucosa specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD patients
  Interventions: Other: no intervention performed- observational only
- Healthy controls
  Interventions: Other: no intervention performed- observational only

INTERVENTIONS:
Other: no intervention performed- observational only — no intervention performed- observational only

SUMMARY:
patients 6-25 years old upon diagnostic evaluation will be recruited . study population will comprise of two groups: newly diagnosed IBD patients/ Celiac disease and healthy controls.

upon enrollment, subjects will fill out sleeping habits questioners, demographic data, medical history.

blood samples will be drawn for CRP and clock gene expression in systemic WBC. intestinal biopsies will be snap frozen for clock gene extraction and amplification only for patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

* IBD or celiac patients with a confirmed diagnosis, recruited upon diagnosis.
* Both male and female
* Age 6-25 years
* Medically treated for IBD in our institute.

Exclusion Criteria:

* Genetic disorder.
* Known primary or secondary immunodeficiency .
* Pregnancy or lactating

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients medically treated in our institute.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
clock gene expression levels in intestinal mucosal samples and WBC peripheral blood. | 4 years
  PCR amplification levels

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Weintraub Y, Cohen S, Yerushalmy-Feler A, Chapnik N, Tsameret S, Anafy A, Damari E, Ben-Tov A, Shamir R, Froy O. Circadian clock gene disruption in white blood cells of patients with celiac disease. Biochimie. 2024 Apr;219:51-54. doi: 10.1016/j.biochi.2023.07.020. Epub 2023 Jul 29. PMID 37524198
- [Derived] Weintraub Y, Cohen S, Anafy A, Chapnik N, Tsameret S, Ben-Tov A, Yerushalmy-Feler A, Dotan I, Tauman R, Froy O. Inverse Relationship Between Clock Gene Expression and Inflammatory Markers in Ulcerative Colitis Patients Undergoing Remission. Dig Dis Sci. 2023 Jun;68(6):2454-2462. doi: 10.1007/s10620-023-07847-y. Epub 2023 Feb 6. PMID 36745299
- [Derived] Weintraub Y, Cohen S, Chapnik N, Ben-Tov A, Yerushalmy-Feler A, Dotan I, Tauman R, Froy O. Clock Gene Disruption Is an Initial Manifestation of Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2020 Jan;18(1):115-122.e1. doi: 10.1016/j.cgh.2019.04.013. Epub 2019 Apr 10. PMID 30981000